CLINICAL TRIAL: NCT02083913
Title: Feasibility and Impacts of a Prebariatric Surgery Exercise Training in Telehealth: a Pilot Study
Brief Title: Prebariatric Surgery Physical Exercise Training in Telehealth
Acronym: TelePreSET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 13-209
Record Dates: First submitted 2014-03-04; First posted 2014-03-11 (Estimated); Last update posted 2018-10-15 (Actual); Status verified 2017-10

CONDITIONS: Obesity
Keywords: Severely obese; Bariatric surgery; Physical activity; Physical fitness; Telehealth; Quality of life
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Supervised physical activity (Experimental)
  Interventions: Behavioral: Telehealth supervised exercise training

INTERVENTIONS:
Behavioral: Telehealth supervised exercise training — Endurance and strength training (3x/week during 12 weeks)

SUMMARY:
The aim of our study is to evaluate the feasibility of a supervised training session using telehealth in the "Clinique medico-chirurgicale du traitement de l'obésité de Sherbrooke" (CMCTO) and its impact on health, physical fitness, quality of life and satisfaction of subjects. 6 subjects awaiting bariatric surgery will be recruited. In addition to usual care, subjects will perform additional sessions of supervised endurance and resistance exercise training. Subjects will be instructed to perform two supervised exercise sessions per week with telehealth plus one without supervision during 12 weeks. The following outcomes will be assessed before and after the telePreSET, then 12 months after bariatric surgery: 1- physical fitness (6MWT, maximal strength, symptom-limited cardiac exercise test); 2-health related quality of life (Laval questionnaire); 3-weight, height, body composition (bioelectrical impedance scale); 4-comorbidities and metabolic parameters (files and blood samples); 5-exercise beliefs (Physical Exercise Belief questionnaire); 6-physical activity (GPAQuestionnaire and actimeter). The feasibility will be assessed with a satisfaction questionnaire concerning physical activity management, dropout and compliance rates, as well as the number of injuries and accidents. The results of this research will give us preliminary data for future projects in order to improve support of bariatric surgery candidates to assure optimal results for their health. Also, we will contribute to the advancement of scientific knowledge, absent in the current literature in this population.

DETAILED DESCRIPTION:
Background: Obesity class II and III increased most rapidly over the past 25 years in Canada and USA. This alarming situation has significantly increased the number of bariatric surgeries performed in North America (101,645 surgeries in 2011). Indeed, bariatric surgery has demonstrated its long-term efficacy in maintaining significant weight loss and in lowering mortality, while reducing the health-care costs of obesity. Unfortunately, bariatric surgery does not always present optimal results in terms of weight loss and resolution of comorbidities, and may be the cause of perioperative complications. The effectiveness of bariatric surgery and the number of perioperative complications are influenced by various factors such as initial weight or physical fitness/activity. For this reasons, various experts recommend regular physical activity in order to optimize the results of bariatric surgery and to decrease perioperative morbidity. However, no interventional studies including pre-surgery exercise training is available in the literature. Preliminary results showed that a supervised Pre-Surgical Exercise Training (PreSET) is feasible and improved physical fitness and quality of life and decreased embarrassment during exercise (Baillot et al. 2013). However, 71.3 % (n = 57) of patients who refused to participate in PreSET explain their refusal because of their schedule, reduced mobility or distance from the hospital. Telehealth is growing and often used for the rehabilitation of cardiac and pulmonary patients. Indeed, it allows to provide equal access to care for people who are geographically remote and are physically and economically disadvantaged. Studies showed that telehealth improve the quality of health care, and may be as effective as face to face meetings to improve the health of patients. The recent decrease in costs related to the equipment makes this intervention modality more accessible. However, no study is available in subjects awaiting bariatric surgery.

Hypothesis and Objectives: Investigators hypothesize that a Telehealth Pre-Surgical Exercise Training (telePreSET) is feasible and will improve the health, physical fitness, quality of life, compliance and satisfaction of subjects. The aim of our study is to evaluate the feasibility in the "Clinique medico-chirurgicale du traitement de l'obésité de Sherbrooke" (CMCTO) of the telePreSET and its impact on health, physical fitness, quality of life and satisfaction of subjects.

Method: 6 subjects awaiting bariatric surgery will be recruited. In addition to usual care, subjects will perform before bariatric surgery additional sessions of supervised endurance and resistance exercise training. Subjects will be instructed to perform two supervised exercise sessions per week with telehealth plus one without supervision during 12 weeks. The following outcomes will be assessed in the different groups before and after the telePreSET, then 12 months after bariatric surgery: 1- physical fitness (6MWT, maximal strength, symptom-limited cardiac exercise test); 2-health related quality of life (Laval questionnaire); 3-weight, height, body composition (bioelectrical impedance scale); 4-comorbidities and metabolic parameters (files and blood samples); 5-exercise beliefs (Physical Exercise Belief questionnaire); 6-physical activity (GPA Questionnaire and actimeter). The feasibility will be assessed with a satisfaction questionnaire concerning PA management, dropout and compliance rates, as well as the number of injuries and accidents.

Issue: The results of this research will give us preliminary data for future projects in order to improve support for bariatric surgery candidates to assure optimal results for their health. Also, we will contribute to the advancement of scientific knowledge, absent in the current literature in this population.

ELIGIBILITY:
Inclusion Criteria:

* bariatric surgery candidate : morbid obesity (BMI>40)or severe obesity (BMI>35 with complications; > 18 years old)
* follow usual care in the "Clinique médico-chirurgicale du traitement de l'obésité du Centre Hospitalier Universitaire de Sherbrooke (CHUS)" and ready to do pre-surgery evaluation (approximately 3 month before surgery)
* no more than one supervised exercise training per week
* inability to come regularly to the CHUS to participate in supervised exercise training
* sufficient space to train at home (4m2)

Exclusion Criteria:

* medical contraindication for physical activity
* major functional limitations: failure to realize the 6 minutes walking test
* intellectual disability and / or neuropsychological disease
* not being able to speak or understand french

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2014-02; Primary Completion 2015-06 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Changes in physical fitness | baseline, then 12 weeks after exercise training and one year after surgery
  6-minutes walking test distance (meter) treadmill symptom-limited cardiac exercise test (METs)

SECONDARY OUTCOMES:
Changes in quality of life scores | baseline, then 12 weeks after exercise training and one year after surgery
  Laval questionnaire
Changes in energy expenditure | baseline, then 12 weeks after exercise training and one year after surgery
  Frequency of subjects reaching 150 min of moderate physical activity Total energy expenditure (kcal per day) Number of steps With accelerometer and international physical activity questionnaire
Changes in weight (kg) | baseline, then 12 weeks after exercise training and one year after surgery
Changes in exercise beliefs | baseline, then 12 weeks after exercise training and one year after surgery
  Exercise beliefs questionnaire: embarrassement, fear of injury, confidence, beliefs in physical activity benefits
Final satisfaction | 12 weeks after exercise training
  Heath care satisfaction questionnaire (% of subjects satisfied + mean score) TeleHeath care satisfaction questionnaire (% of subjects satisfied + mean score)
Changes in body composition | aseline, then 12 weeks after exercise training and one year after surgery
  % of fat mass and fat free mass (bioimpedancemeter)
Changes in comorbidities | baseline, then 12 weeks after exercise training and one year after surgery
  Medical charts: % of subjects with diabetes, hypertension, dyslipidemia, sleep apnea, depression, anxiety, arthrosis, osteoarthrosis
Final compliance | 12 weeks after the beginning of the intervention
  Adherence of sessions Number of injuries or adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Marie-France Langlois, MD, Principal Investigator — Université de Sherbrooke
Locations (1):
- Centre hospitalier universitaire de Sherbrooke, Sherbrooke, Quebec, Canada

REFERENCES:
- [Background] Baillot A, Mampuya WM, Comeau E, Meziat-Burdin A, Langlois MF. Feasibility and impacts of supervised exercise training in subjects with obesity awaiting bariatric surgery: a pilot study. Obes Surg. 2013 Jul;23(7):882-91. doi: 10.1007/s11695-013-0875-5. PMID 23430477